CLINICAL TRIAL: NCT01198652
Title: Belfort Dildy- Obstetrical Tamponade System Post-Marketing Surveillance Program
Status: Terminated | Type: Observational
Why Stopped: Study discontinued following 57 subjects enrolled over 2 years
Sponsor: Glenveigh Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 04
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Postpartum Uterine Bleeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Belfort-Dildy Obstetric Tamponade Tx: Patients treated with Belfort-Dildy Obstetric Tamponade System are eligible for inclusion in the cohort.

SUMMARY:
This is an open, post-marketing surveillance study obtaining data retrospectively on 300 women, of any age, treated with the BD-OTS for postpartum uterine bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with the BD-OTS device

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received treatment with the BD-OTS as part of their standard of care in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Adair, MD, Study Director — Glenveigh Medical
Locations (11):
- United States (11):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Presbyterian/St. Luke's Medical Center, Denver, Colorado
  - Orlando Health, Orlando, Florida
  - Monmouth Medical Center, Long Branch, New Jersey
  - UHS - Wilson Medical Center, Johnson City, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Erlanger, Chattanooga, Tennessee
  - St. David's Medical Center, Austin, Texas
  - North Austin Medical Center - St. David's Women's Center of Texas, Austin, Texas